CLINICAL TRIAL: NCT07294313
Title: Harnessing Artificial Intelligence for Diagnosing Androgenetic Alopecia: A Training and Validation Study
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noura Adel Ahmed Abdelghany Nour, Assistant Lecturer, Cairo University
Other Study IDs: MD-192-2025
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Androgenetic Alopecia
Keywords: Androgenetic Alopecia; deep learning; Artificial Intelligence; Convoluted neural network; trichoscopy; female pattern hair loss; male pattern hair loss; handheld dermoscope; hair count
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- androgenetic alopecia: Patients diagnosed clinically and trichoscopically with androgenetic alopecia of both genders. The diagnosis of AGA requires fulfillment of the primary criterion, plus one or more of the secondary criteria, and absence of exclusion criteria:
  * Primary criterion Hair shaft thickness heterogeneity on the frontal and/or vertex scalp, defined as proportion of hairs < 0.06 mm (including intermediate, thin, and vellus hairs) ≥20%.
  * Secondary criteria
    1. Proportion of single hair follicle unit on the frontal and/or vertex scalp ≥30%.
    2. Proportion of vellus hairs on the frontal and/or vertex scalp >10%.
    3. There are at least two other dermoscopic signs: brown peripilar sign, yellow dots,white dots, scalp honeycomb pigmentation
  * Exclusion criteria Black dots, broken hairs, exclamation mark hairs
- normal controls: apparently normal participants not suffering from the following :
  1. androgenetic alopecia
  2. patchy hair loss.
  3. cicatricial alopecia or diffuse alopecia areata
  4. inflammatory scalp disorders (psoriasis, seborrheic dermatitis, lichen planopilaris and frontal fibrosing alopecia in a pattern distribution)

SUMMARY:
The aim of this study is to develop and validate deep learning models in diagnosis of male and female pattern hair loss, and assessment of its severity based on clinical and trichoscopic image by handheld dermoscopy and administrative data (age and sex).

DETAILED DESCRIPTION:
The investigators intend to develop and validate artificial intelligence (AI) and machine learning (ML) models in diagnosis of male and female pattern hair loss, and assessment of its severity based on clinical and trichoscopic image using widely available and accessible handheld dermoscopes.

Conventional androgenetic alopecia (AGA) diagnosis and severity assessment are tedious and time-consuming tasks that are prone to human errors. These challenges can be tackled using artificial intelligence (AI), namely leveraging applications of machine learning and artificial neural networks for enhancing the diagnostic accuracy of scalp disease classification systems via dermoscopic image analysis. Computer aided assessment of hair microphotographs was attempted for decades, yet it faced many technical hurdles before the onset of deep learning and neural networks; and currently available software generate inaccurate results compared with visual counting. More accurate methods of analysis are needed for trichoscopic imaging, utilising deep learning image recognition models trained with a large image dataset. A number of deep learning models have been developed in recent years using videodermoscopy that achieved reliable hair density, thickness and severity classification, yet remain limited by small non-inclusive training datasets, need for hair shaving and lack of detailed reporting. Moreover, to our knowledge all previous models depend on image acquisition from expensive standalone videodermoscopy devices that lack widespread availability, rather than handheld dermoscopes that are commonly available.

The study will enroll 400 participants (200 healthy controls and 200 AGA patients). Controls undergo history and trichoscopic exams to exclude hair disorders. Trichoscopic examination will be conducted using a handheld dermoscope (CuTechs DS175) with a specialized field spacer. Patients will be assessed for disease severity using gender-specific scales. Both groups will have standardized digital and trichoscopic images taken for analysis. Images will be used to manually count and classify hairs, assess follicle units, and identify dermoscopic signs. A structured database will store all data and link clinical and image data to support objective diagnosis. AI models, particularly CNNs using transfer learning, will be trained on preprocessed images for classification and severity scoring. Model performance will be evaluated using metrics like accuracy, precision, recall, F1-score, and AUC-ROC compared with metrics reported by expert trichologists to validate accuracy and reliability

ELIGIBILITY:
for the patient group:

Inclusion criteria:

* Patients with male or female pattern hair loss diagnosed clinically or suspected clinically and confirmed trichoscopically
* Age of disease onset 12-50 years old
* Both genders
* Any grade of androgenetic alopecia
* Any duration of androgenetic alopecia
* Any skin type

Exclusion criteria by clinical and trichoscopic examination:

* Patients with patchy hair loss or Telogen effluvium only.
* Patients with cicatricial alopecia or diffuse alopecia areata
* Patients with inflammatory scalp disorders (psoriasis, seborrheic dermatitis, lichen planopilaris and frontal fibrosing alopecia in a pattern distribution)
* Lack of patient cooperation.

for the control group: apparently healthy participants not suffering from the following: AGA, patchy hair loss, cicatricial alopecia, diffuse alopecia areata, inflammatory scalp disorders (psoriasis, seborrheic dermatitis, lichen planopilaris and frontal fibrosing alopecia in a pattern distribution).

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients diagnosed clinically and trichoscopically with androgenetic alopecia of both genders and apparently healthy controls.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
assessment of diagnostic capability of AI in AGA | 1 year
  Assess accuracy, sensitivity, specificity and positive predictive value of the trained AI models in differentiating AGA affected from non-AGA affected subjects using their macroscopic and trichoscopic images.

SECONDARY OUTCOMES:
assessment of severity of androgenetic alopecia using AI | 1 year
  Assess accuracy, sensitivity, specificity and positive predictive value of the trained AI models in assessment of severity of androgenetic alopecia as regards:
  1. Clinical classification (Sinclair scale for female pattern baldness and the Hamilton-Norwood scale for male pattern baldness)
  2. Trichoscopic parameters: mean hair thickness (in micrometer, using planimetric analysis), hair density (frequency per cm2), proportion of terminal hairs, proportion of vellus hairs, number of hairs per follicular unit, presence of brown peripilar sign, yellow dots, and scalp honeycomb pigmentation.
facilitation of AI assessment using macroscopic imagies | 1 year
  To compare the model's diagnostic accuracy using the macroscopic versus trichoscopic images alone

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
relevant praticipant data shall be provided to researchers who request them on reasonable basis
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from 2027 indefintely
Access Criteria: access will be provided to deidentified data including all study parameters

REFERENCES:
- [Background] Sacha JP, Caterino TL, Fisher BK, Carr GJ, Youngquist RS, D'Alessandro BM, Melione A, Canfield D, Bergfeld WF, Piliang MP, Kainkaryam R, Davis MG. Development and qualification of a machine learning algorithm for automated hair counting. Int J Cosmet Sci. 2021 Nov;43 Suppl 1:S34-S41. doi: 10.1111/ics.12735. PMID 34426987
- [Background] Wang Y, Ding W, Yao M, Li Y, Wang M, Wang L, Li Z, Sun S, Yang M, Zhu Y, Zhou N. Diagnostic and grading criteria for androgenetic alopecia using dermoscopy. Skin Res Technol. 2024 Apr;30(4):e13649. doi: 10.1111/srt.13649. PMID 38533753
- [Background] Kuczara A, Waskiel-Burnat A, Rakowska A, Olszewska M, Rudnicka L. Trichoscopy of Androgenetic Alopecia: A Systematic Review. J Clin Med. 2024 Mar 28;13(7):1962. doi: 10.3390/jcm13071962. PMID 38610726
- [Background] Young AT, Xiong M, Pfau J, Keiser MJ, Wei ML. Artificial Intelligence in Dermatology: A Primer. J Invest Dermatol. 2020 Aug;140(8):1504-1512. doi: 10.1016/j.jid.2020.02.026. Epub 2020 Mar 27. PMID 32229141
- [Background] Devjani S, Ezemma O, Kelley KJ, Stratton E, Senna M. Androgenetic Alopecia: Therapy Update. Drugs. 2023 Jun;83(8):701-715. doi: 10.1007/s40265-023-01880-x. Epub 2023 May 11. PMID 37166619
- [Background] Bokhari L, Cottle P, Grimalt R, Kasprzak M, Sicinska J, Sinclair R, Tosti A. Efficiency of Hair Detection in Hair-to-Hair Matched Trichoscopy. Skin Appendage Disord. 2022 Sep;8(5):382-388. doi: 10.1159/000524345. Epub 2022 May 12. PMID 36161091